CLINICAL TRIAL: NCT04172493
Title: Hyperspectral Endoscopy Imaging for Early Detection of Precancerous Lesions in Average Risk Patients: Proof of Principle
Brief Title: Hyperspectral Endoscopy Imaging for the Early Detection of Precancerous Lesions in Average Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Vassiliki Tsikitis, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00018947; NCI-2019-06087 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ONC-19132-L; STUDY00018947 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-21 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Patient

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diagnostic (Experimental): Patients undergo standard of care white light endoscopy (WLE) and hyperspectral endoscopy (HySE) during routine colonoscopy procedure.
  Interventions: Procedure: Hyperspectral Endoscopy (HySE); Device: White Light Endoscopy (WLE)

INTERVENTIONS:
Procedure: Hyperspectral Endoscopy (HySE) — Undergo hyperspectral endoscopy
  Other Names: Hyperspectral Endoscopic Imaging (HSI)
Device: White Light Endoscopy (WLE) — Undergo white light endoscopy
  Other Names: White Light Endoscopic Imaging

SUMMARY:
This trial studies whether hyperspectral endoscopy improves visualization of abnormal tissue in average risk patients during standard-of-care colonoscopies. Hyperspectral endoscopy is an emerging technique that has the potential to enable the signals from blood to be resolved from tissue-specific signals. Image-enhanced endoscopy may improve visualization of abnormal colonic tissue when compared to the standard-of-care high-definition white light endoscopy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess whether use of hyperspectral endoscopy (HySE) can improve visualization of abnormal colonic tissue.

SECONDARY OBJECTIVES:

I. To assess whether use of HySE could reduce the rate of missed flat polyps.

II. To assess whether use of HySE might in the future reduce the incomplete resection rate (IRR).

III. To examine accuracy of practitioners in predicting polyp histology.

OUTLINE:

Patients undergo standard of care white light endoscopy and hyperspectral endoscopy during routine colonoscopy procedure.

After completion of study, patients who experience a colonoscopy-related severe adverse event are followed up until resolution or stabilization of the event.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Patients scheduled for a standard of care screening or surveillance colonoscopy

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, precludes the patient from completion of the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Spectral profiles corresponding to normal versus abnormal colonic tissue | 1 year
  Will apply a multivariate statistical analysis such as spectral angle mapper to determine whether the spectra are significantly different as determined by light spectral bandwidth measurements.
Image quality | 1 year
  Assessed by the endoscopist, based on level of confidence in delineating the area of interest. Will assess and compare the number of polyps found by standard light endoscopy and narrow band imaging with hyperspectral endoscopy.

SECONDARY OUTCOMES:
Imaging differences in polyp characteristics documented upon post-procedure video review | 1 year
  Will be compared with the final read of the pathology of the polyps. A Pearson X2 test or equivalent test will be applied. When applicable, Fisher exact test and Pearson X2 test will be used to test for differences in categorical variables, which include analysis of polyp morphologic structure and location. A student t test or equivalent statistical test will be used to test for differences in continuous variables, including polyp diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki L Tsikitis, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States